CLINICAL TRIAL: NCT06265688
Title: An Investigational Study of CX-2051 in Participants With Advanced Solid Tumors
Brief Title: First In Human Study of CX-2051 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CytomX Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMX-2051-101
Record Dates: First submitted 2024-02-12; First posted 2024-02-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Solid Tumor, Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CX-2051 (Experimental)
  Interventions: Drug: CX-2051

INTERVENTIONS:
Drug: CX-2051 — Investigational drug monotherapy

SUMMARY:
The purpose of this first-in-human study, CTMX-2051-101, is to characterize the safety, tolerability, and antitumor activity of CX-2051 in adult participants with advanced solid tumors.

DETAILED DESCRIPTION:
The study is comprised of 2 parts. Part 1 involves CX-2051 dose escalation to identify the maximum tolerated dose (MTD) of CX-2051. Part 2 (dose expansion) will further assess safety and tolerability as well as preliminarily assess antitumor activity of CX-2051 in indication-specific expansion cohorts.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced unresectable solid tumor that has progressed after standard therapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Measurable disease per RECIST v1.1
* Consent to fresh biopsy or if medically contraindicated, recent (within 6 months) archival tumor tissue
* Additional inclusion criteria may apply

Exclusion Criteria:

* Recent history (within last 2 years) of localized cancers that are not related to the current cancer being treated
* Known active central nervous system (CNS) involvement by malignancy
* Systemic anticancer treatment, radiotherapy, or investigational agent(s) within 14 days prior to C1D1
* Previous treatment with antibody-drug conjugates (ADCs) with Topo-I inhibitor payload
* Major surgery (requiring general anesthesia) within 4 weeks prior to C1D1
* Elevated baseline laboratory values
* Serious concurrent illness
* Pregnant or breast feeding
* Additional exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2029-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of CX-2051 | 44 months
  The number of participants experiencing a dose-limiting toxicity (DLT) as defined in the protocol, AEs (adverse events), and treatment-emergent adverse events (TEAEs) at any dose level
Determine the recommended Phase 2 dose (RP2D) | 44 months
  The number of participants experiencing a dose-limiting toxicity (DLT) as defined in the protocol, AEs (adverse events), and treatment-emergent adverse events (TEAEs) at any dose level

SECONDARY OUTCOMES:
Objective response rate (ORR) | 60 months
  ORR defined as the proportion of participants who achieve a confirmed complete response (CR) or partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Investigator assessment
Duration of response (DOR) | 60 months
  DOR defined as the time from the first documentation of confirmed CR or PR (based on RECIST v1.1) to the first documentation of disease progression or death due to any cause on study, whichever occurs first.
Progression-free survival (PFS) | 60 months
  PFS defined as the time from the first dose of study intervention to the date of first documentation of objective tumor progression (based on RECIST v1.1) or death due to any cause, whichever occurs first.
Disease control rate (DCR) | 60 months
  DCR defined as the proportion of participants with confirmed CR, PR, or stable disease (SD) as per RECIST v1.1 by Investigator assessment.
Duration of disease control (DODC) | 60 months
  DODC defined as the time from the first documentation of confirmed CR, PR, or SD (based on RECIST v1.1) to the first documentation of disease progression or death due to any cause on study, whichever occurs first.
Overall survival (OS) | 60 months
  OS defined as the time from the first dose of study intervention to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Monika Vainorius, MD, Study Director — CytomX Therapeutics
Locations (4):
- United States (4):
  - Sarah Cannon Research Institute at HealthONE, Denver, Colorado
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Carolina BioOncology Institute, PLLC, Huntersville, North Carolina
  - Sarah Cannon Research Institute, LLC, Nashville, Tennessee